CLINICAL TRIAL: NCT01653587
Title: Randomized Trial Between the Transfemoral Approach With AngioSeal and the Transradial Approach to Prevent Vascular Access Complications in Non-ST-Segment Elevation Acute Coronary Syndrome Patients Submitted To Early Invasive Strategy
Brief Title: AngioSeal Versus Radial Approach in Acute Coronary Syndrome
Acronym: ARISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Irmandade Santa Casa Misericórdia Marília (Other)
Responsible Party: Principal Investigator, Pedro Beraldo de Andrade, MD, Irmandade Santa Casa Misericórdia Marília
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ISCMM-01; PBA-1 (Other: ISCMM-PBA)
Record Dates: First submitted 2012-07-26; First posted 2012-07-31 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Transradial Approach; Transfemoral Approach; Vascular Closure Device
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transradial approach (Active Comparator): Transradial approach percutaneous coronary intervention using the TR Band device to obtain hemostasis
  Interventions: Device: Percutaneous coronary intervention
- Transfemoral approach (Active Comparator): Transfemoral approach percutaneous coronary intervention using the AngioSeal vascular closure device STS Plus Platform to obtain hemostasis
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — Both transradial and transfemoral coronary angiography will be performed by the Judkins technique using arterial introducers with 6 French diameter and pre-molded catheters for selective catheterization of left and right coronary arteries.Percutaneous coronary intervention will be indicated when a culprit lesion is identified, with stenosis diameter severity ≥ 70%, with high probability of angiographic success, being ideally performed immediately after coronary angiography and left ventriculography. Patients with multiarterial coronary disease will be submitted to percutaneous coronary intervention after agreement among cardiologist, interventional cardiologist and thoracic surgeon. Procedures will be performed according to recommendations and provisions of current guidelines.
  Other Names: AngioSeal vascular closure device; TR Band radial artery compression device

SUMMARY:
Among non-ST-segment elevation acute coronary syndrome patients submitted to early invasive strategy and randomized for the transfemoral or transradial approach, the AngioSeal vascular closure device would decrease the prevalence of vascular complications at puncture site, reaching the non-inferiority criterion when compared to the radial access.

DETAILED DESCRIPTION:
Antithrombotic therapy and percutaneous or surgical myocardial revascularization procedures are the basis of the treatment of patients admitted with non-ST-segment elevation acute coronary syndrome. However, the desired reduction of the recurrence of ischemic events has as complication an increased incidence of bleeding. Since arterial puncture followed by the insertion of an introducer has become the standard method to perform invasive cardiovascular procedures, complications related to vascular access have become an important bleeding site.

Among the strategies to decrease vascular complications, the transradial approach is a well stablished alternative to the transfemoral approach. For its part, vascular closure devices were introduced to decrease vascular complications, homeostasis time and ambulation time of patients submitted to invasive procedures by the transfemoral access. Rapidly incorporated to the clinical practice, such devices to date have shown conflicting results with regard to their safety and efficacy. The inconsistency of data proving its safety limits its routine adoption as strategy to prevent vascular complications, requiring evidences through adequately designed randomized studies for this end.

ELIGIBILITY:
Inclusion Criteria:

* Non-ST-segment elevation ACS patients [ischemic symptoms suspicious of non-ST-segment elevation ACS (unstable angina or non-ST-segment elevation AMI) defined as clinical presentation compatible with a new manifestation of worsening of chest pain characteristic of ischemia, at rest or at minimum effort, lasting more than 10 minutes, and at least one of the following items: (a) ECG changes compatible with new ischemia (ST segment depression of at least 1 mm, or transient ST segment elevation, or ST segment elevation ≤ 1 mm, or T wave inversion > 2 mm in at least 2 contiguous shunts); (b) cardiac enzymes (CK-MB or troponin T or I) above the upper normality range limit; (c) patients > 60 years of age without ECG or myocardial necrosis markers changes, however with previous documentation of coronary atherosclerotic disease (CAD), confirmed by previous hospitalization due to AMI, previous percutaneous or surgical myocardial revascularization procedure, significant CAD confirmed by coronary angiography, or positive functional test for myocardial ischemia];
* Intention to submit patient to early invasive strategy consisting of coronary angiography immediately followed by PCI, when applicable, in the first 72 hours after admission;
* Signed informed consent;
* Patient eligible for transradial and transfemoral coronary angiography and PCI, being pre-requisites: (a) palpable radial artery with normal Allen test or/and oximetry tests, (b) familiarity of the operator with the radial and femoral techniques using AngioSeal, (c) agreement of the operator to use the access route determined by the randomization process.

Exclusion Criteria:

* Less than 18 years of age;
* Pregnancy;
* Chronic use of vitamin K antagonists or direct thrombin inhibitors, or oral Xa-factor antagonists;
* Hypersensitivity to antiplatelet and/or anticoagulant drugs;
* Active bleeding or high bleeding risk (severe liver failure, active peptic ulcer, creatinine clearance < 30 mL/min, platelets count < 100.000 mm3);
* Uncontrolled systemic hypertension;
* Cardiogenic shock;
* Previous myocardial revascularization surgery with ≥ 1 internal mammary or radial artery graft;
* Documented chronic peripheral arterial disease preventing the use of the femoral technique;
* Severe concomitant disease with life expectancy below 12 months;
* Participation in drug or devices investigative clinical trials in the last 30 days;
* Indication of elective percutaneous coronary intervention to be performed in a moment different from immediately after coronary angiography;
* Medical, geographic or social conditions impairing the participation in the study or inability to understand and sign the informed consent term.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro B Andrade, MD, Principal Investigator — Irmandade da Santa Casa de Misericórdia de Marília
Locations (1):
- Irmandade da Santa Casa de Misericórdia de Marília, Marília, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Andrade PB, E Mattos LA, Tebet MA, Rinaldi FS, Esteves VC, Nogueira EF, Franca JI, de Andrade MV, Barbosa RA, Labrunie A, Abizaid AA, Sousa AG. Design and rationale of the AngioSeal versus the Radial approach In acute coronary SyndromE (ARISE) trial: a randomized comparison of a vascular closure device versus the radial approach to prevent vascular access site complications in non-ST-segment elevation acute coronary syndrome patients. Trials. 2013 Dec 18;14:435. doi: 10.1186/1745-6215-14-435. PMID 24345099
- [Result] Andrade PB, Mattos LA, Rinaldi FS, Bienert IC, Barbosa RA, Labrunie A, Tebet M, Esteves V, Abizaid A, Sousa AR. Comparison of a vascular closure device versus the radial approach to reduce access site complications in non-ST-segment elevation acute coronary syndrome patients: The angio-seal versus the radial approach in acute coronary syndrome trial. Catheter Cardiovasc Interv. 2017 May;89(6):976-982. doi: 10.1002/ccd.26689. Epub 2016 Aug 12. PMID 27514319

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transradial Approach | Transfemoral Approach
Started | 120 | 120
Completed | 120 | 120
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transradial Approach | Transfemoral Approach | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 67 | 132
  >=65 years | 55 | 53 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (11.2) | 63.6 (10.2) | 63.0 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 24 | 64
  Male | 80 | 96 | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 120 | 120 | 240
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 120 | 120 | 240
Region of Enrollment [Number; unit: participants]
  Brazil | 120 | 120 | 240

OUTCOME MEASURES:

1. Primary Outcome: First Occurrence of Access Site Related Ischemic or Bleeding Complication
Description: Vascular and systemic complications at arterial puncture site include major bleeding, retroperitoneal hemorrhage, compartment syndrome, hematoma ≥ 5 cm, pseudoaneurysm, arteriovenous fistula, infection, limb ischemia, asymptomatic arterial occlusion, adjacent nerve injury or need for vascular surgery repair.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Transradial Approach | Transfemoral Approach
Number analyzed (Participants) | 120 | 120
Participants | 16 | 15

2. Secondary Outcome: Adverse Ischemic or Bleeding Events
Description: Individual components of the primary objective, hematoma < 5 cm, cardiovascular death, myocardial infarction, stroke, major bleeding unrelated to puncture site or to coronary artery bypass grafting, device success and crossover rate between techniques
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Transradial Approach | Transfemoral Approach
Number analyzed (Participants) | 120 | 120
Participants | 11 | 3

3. Other Pre Specified Outcome: Cardiovascular Death, Myocardial Infarction or Stroke
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Transradial Approach | Transfemoral Approach
Number analyzed (Participants) | 120 | 120
Participants | 2 | 3

ADVERSE EVENTS:
Arm/Group | Transradial Approach | Transfemoral Approach
All-Cause Mortality (participants affected / at risk) | 2/120 | 2/120
Serious Adverse Events (participants affected / at risk) | 3/120 | 9/120
Other Adverse Events (participants affected / at risk) | 2/120 | 2/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transradial Approach (N=120) | Transfemoral Approach (N=120)
Cardiovascular death (Cardiac disorders) | 0 (0) | 2 (2)
Total mortality (General disorders) | 1 (1) | 2 (2)
Periprocedural myocardial infarction (Cardiac disorders) | 2 (2) | 4 (4)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transradial Approach (N=120) | Transfemoral Approach (N=120)
Major bleeding (Vascular disorders) | 2 (2) | 2 (2) — Type 3 or 5 according to BARC definition

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No